CLINICAL TRIAL: NCT03703232
Title: An Adaptable Foot Prosthesis for People With Lower Extremity Amputations - Community Experiences
Brief Title: Community Walking Trials: Comparing Prosthetic Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: WillowWood Global LLC (Industry)
Responsible Party: Principal Investigator, Murray Maitland, Associate Professor, School of Medicine, Rehabilitation Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00001109
Record Dates: First submitted 2018-04-03; First posted 2018-10-11 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: Lower Extremity Amputation
Keywords: prosthesis; prosthetic; foot; ankle; mobility; amputee

STUDY DESIGN:
Intervention Model Description: The research design is an A-B-A design, where the A condition is the participant's usual prosthetic foot and the B condition is the investigational foot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lower extremity amputees (Other): Community walking trial comparing usual prosthetic foot with investigational prosthetic foot.
  Interventions: Device: Investigational prosthetic foot

INTERVENTIONS:
Device: Investigational prosthetic foot — Individuals will complete 2-4 weeks of community walking with the investigational foot and compare to their regular prosthetic foot.

SUMMARY:
The purpose of the study is to obtain performance measurements and participant feedback about use of an investigational prosthetic foot compared to the participant's usual prosthetic foot. To accomplish this, the study will use a combination of laboratory motion analysis, functional tests, and community mobility trials where participants complete questionnaires and interviews about use of an investigational prosthetic foot compared to the participant's usual prosthetic foot.

Individuals with amputations that participate in the (optional) motion analysis sub-study at the University of Washington will complete forward walking, side-step, and across river rock with usual foot (session 1), and also with the investigational foot locked and unlocked (session 2) after an accommodation period of between 1-4 weeks. The participants will rate their experiences using socket comfort score and the socket pressure score.

Control participants recruited at the University of Washington to provide information about performance for people without amputation will go through the consenting process, then will be asked to complete forward walking, Figure-of-8 Walk Test, Narrowing Beam Walking Test, side-step, and walking across river rock surface. These tests will be conducted at a single session.

DETAILED DESCRIPTION:
If the participant with an amputation is eligible and wishes to participate, an appointment will be made for the person to come to the University of Washington Motion Analysis Lab or WillowWood, in Mt. Sterling, Ohio. The participant will meet with a researcher and clinical prosthetist to go through the consenting process. At that time, participants will complete the demographic data questionnaire.

The prosthetist will assess the condition and fit of the participant's current prosthesis for alignment, fit, and condition. The prosthetist will also inspect the participant's residual limb for skin condition. People presenting with significant skin breakdown will not be eligible to participate. The prosthetist will also determine how best to set up the current socket system with the investigational foot at that time.

Motion analysis trials of the investigational foot compared to the participant's usual foot. Participants will complete forward walking, side-step, and across river rock with usual foot (session 1), and also with the investigational foot locked and unlocked (session 2) after an accommodation period of between 1-4 weeks. The UW will conduct optically-based motion analysis using an 8-camera Qualisys motion capture system 4 embedded tri-axial ground reaction force platforms and a river rock-substrate surface that is parallel to the main motion capture space. For all motion analysis tests, retroreflective markers are taped to anatomical landmarks that are compatible with Visual 3-D kinematic modeling software. Motion data are captured at 120 Hz.

Motion Analysis Tests Forward walking. Participants will walk at a self-selected speed on a level surface for 10 m. In the center of the calibrated walking area, the participant will step on force plates. Marker position and reaction forces will be recorded for 2 sequential steps of the prosthetic side for participants with amputations, or matched side for control subjects. After a practice test, 3 tests where the prosthetic side successfully contacts the force plates will be recorded.

Side-step. Participants will perform the test in a similar manner to forward walking but will instead move laterally over the 10 m surface and across the centrally placed force plates. The order of side-stepping to the right or left will be randomly assigned. Participants will be asked not to cross-over their feet. After a practice test, 3 tests in each direction, where the prosthetic side or matched side successfully contacts the force plates, will be recorded.

Walking across river rock surface. Participants will walk in a direct path through the center of the river rock. They will be wearing a safety harness and will be attached to an overhead moving protection system. Participants will use the visual field limiting goggles during the river rock walking test. After practice tests, 3 tests will be recorded.

Modified socket comfort score and pressure score. Following each test protocol, participants will be asked to rate the socket comfort during the activity from 0 to 10 (with 0 being the least comfortable and 10 being the most comfortable imaginable) and pressures of the prosthetic socket on their residual limb during the activity from 0 to 10 (with zero being none and 10 being the highest imaginable). Participants will be asked to qualify the score with subjective comments.

Community Walking Trials (CWT) of the Investigational foot. To assess the benefit of the investigational foot, a combination of subjective and objective measures will be collected following 2- to 4-week periods of use. During the first laboratory visit, subjects will complete functional tasks with their existing prosthesis, as well as complete the Prosthetic Evaluation Questionnaire (PEQ) and the Comprehensive Lower Limb Amputee Socket Survey (CLASS). Next, they will be fit with the investigational foot and complete a 2- to 4-week at-home use period. A team member will contact the participant about one week after they start using the investigational foot to see how things are going and if there are any issues or problems to address (such as is the degree of stiffness appropriate) that may prompt a re-fitting. If this occurs, the 2- to 4-week at-home use period will re-start, increasing the participant's total amount of time in the study. During at-home use, participants will be prompted to complete a daily, structured, online logbook formatted in REDCap.

During the second visit, subjects will again complete the PEQ and CLASS, and repeat the same functional tasks as at the first visit but while wearing the investigational foot (locked and unlocked linkage). During this visit, a semi-structured interview will be conducted and recorded using Zoom. At the end of the visit, subjects will be re-fit with their original prosthetic foot and will complete another 2- to 4-week at-home use period with logbook entries before completing study questionnaires and a final interview.

Quantitative instruments - Community Walking Trials PEQ Subscales: The PEQ is a 9-scale instrument that has good psychometric properties and has been validated. The PEQ subscales vary from 0 (worst) to 100 (best). PEQ subscales of residual limb health, ambulation, utility, and sounds were selected for this study and comprise a total of 24 visual analogue scale questions.

CLASS: The intent of the CLASS is to provide greater insight into the cause of socket dissatisfaction compared to the Socket Comfort Score. To accomplish this, the CLASS includes 4 subcategories; 1) stability, 2) suspension, 3) comfort, and 4) appearance. Each subcategory contains 3-4 items scored using a 5-point scale that relate to common tasks such as standing, sitting, walking, and ascending and descending stairs.

Semi-structured interview: Participants' lived experiences using the investigational foot in comparison to the participant's usual foot will be collected using qualitative research methods. There will be an exit interview using open-ended questions to obtain qualitative data on foot performance and comparisons of foot prostheses. The interviews will be audio recorded. Interviews may be conducted remotely.

Daily Log Book: During home use of the participant's usual foot and the investigational foot, participants will keep an activity log (completed either electronically or on paper) that encourages descriptions of activities, including strengths and limitations of foot performance.

Functional Tasks Figure-of-8 Walk Test: Subjects will begin the task standing between the 2 cones. The subject will walk a figure-of-8 course 3 times for each condition at their self-selected pace and stop when they return to the start position. Time to complete the test and number of steps will be collected.

Narrowing Beam Walking Test:

The test consists of walking across a beam that has 4, 6-foot long sections, each one narrower than the previous one. The narrowing beam is 2" above the floor. When ready, the subject will begin walking along the beam while keeping their feet pointed in the direction of the beam (no side-stepping allowed). Subjects must keep their arms crossed in front of their body to eliminate the use of their arms to maintain balance. For this test of balance, the distance along the beam will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral below knee amputation, use a prosthetic foot for at least 1 year
* Ability to walk 400 meters on level ground without using a walking aid and without an increase in pain
* Ability to read, write, and comprehend English

Exclusion Criteria:

* Residual skin breakdown
* Weight over 300 lbs

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Maitland, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legro MW, Reiber GD, Smith DG, del Aguila M, Larsen J, Boone D. Prosthesis evaluation questionnaire for persons with lower limb amputations: assessing prosthesis-related quality of life. Arch Phys Med Rehabil. 1998 Aug;79(8):931-8. doi: 10.1016/s0003-9993(98)90090-9. PMID 9710165

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lower Extremity Amputees
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Investigational Foot and Usual Foot in the Prosthetic Evaluation Questionnaire (PEQ): Ambulation Sub-Scale
Description: Self-report questionnaire. PEQ Subscales: The PEQ is a 9-scale instrument that has good psychometric properties and has been validated. The PEQ subscales have a range from 0 (worst) to 100 (best). PEQ subscales of residual limb health, ambulation, utility, and sounds were selected for this study and comprise a total of 24 visual analogue scale questions. ICC estimates for these subscales for the first and second administration ranged from 0.79 to 0.9.
Time Frame: Baseline (A1), after 2-week trial of investigational foot (B), after return to usual foot for 2 weeks (A2). Primary analysis uses B minus A2.
Population: All participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | 4.2 (12.9)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.092, Wilcoxon signed-rank test

2. Primary Outcome: Difference Between Investigational Foot and Usual Foot in the Comprehensive Lower Extremity Amputee Socket Survey (CLASS): Comfort Scale
Description: The intent of the CLASS is to provide greater insight into the cause of socket dissatisfaction compared to the Socket Comfort Score. To accomplish this, the CLASS includes 4 subcategories; 1) stability, 2) suspension, 3) comfort, and 4) appearance. Each subcategory contains 3-4 items scored using a 5-point scale that relate to common tasks such as standing, sitting, walking, and ascending and descending stairs.
  Scale range: 0-60 Values: 0 = worst outcome; 60 = best outcome Subscales:0-16
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | 1.1 (11.6)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.760, Wilcoxon signed-rank test

3. Primary Outcome: Difference Between Investigational Foot and Usual Foot in the Figure-of-8 Walking Test: Time
Description: The F8W was developed to represent walking skills used in everyday life, involving straight and curved paths in both right and left directions. It has been validated in older adult populations with mobility disability. Subjects will begin the task standing between the 2 cones. The subject will walk a figure 8 course 3 times for each condition at their self-selected pace and stop when they return to the start position. The outcomes of the test are the time to complete the course.
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
seconds | -0.53 (1.08)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.007, Wilcoxon signed-rank test

4. Primary Outcome: Difference Between Investigational Foot and Usual Foot in the Daily Activity Log: Scale Measuring How Prosthesis Helps or Hinders When Walking on a Challenging Surface
Description: Difference between investigational foot and usual foot of the average daily values of the visual analog scale of participant's perception of gait on challenging surface.
  Scale range: 0-100 Values: 0 = worst outcome; 100 = best outcome
Time Frame: Daily for 2-4 weeks
Population: All participants with a recorded score for both investigational and usual foot were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 29
score on a scale | 10.5 (17.9)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.003, Wilcoxon signed-rank test

5. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Prosthetic Evaluation Questionnaire (PEQ): Residual Limb Health Subscale
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | 1.6 (12.8)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.861, Wilcoxon signed-rank test

6. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Comprehensive Lower Extremity Amputee Socket Survey (CLASS): Stability Subscale
Description: The intent of the CLASS Stability Subscale is to provide greater insight into the cause of socket dissatisfaction compared to the Socket Comfort Score. This subcategory of the CLASS contains 4 items scored using a 5-point scale that relate to common tasks such as standing, sitting, walking, and ascending and descending stairs.
  Values: 0 = worst outcome; 16 = best outcome
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | 3.2 (10.2)

7. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Narrowing Beam Walking Test: Distance Travelled
Description: The Narrowing Beam Walking Test was developed to measure balance in lower extremity amputees (LEA) and it was validated in LEPU with and without a history of falls. The test consists of walking across a beam that has 4, 6-foot long sections, each one more narrow than the previous one. The narrowing beam is 2" above the floor. Subjects must keep their arms crossed in front of their body to eliminate the use of their arms to maintain balance. The distance of the furthest point of contact from the start of the beam is used as the outcome for the test.
Time Frame: Baseline (A1), after 2-week trial of investigational foot (B). Primary analysis uses B minus A1.
Population: All
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
feet | 0.45 (2.34)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.405, Wilcoxon signed-rank test

8. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Daily Activity Log: Balance Confidence
Description: Difference between investigational foot and usual foot of the average daily values of the visual analog scale of participant's perception of balance confidence.
  Scale range: 0-100 Values: 0 = worst outcome; 100 = best outcome
Time Frame: Average of daily measurements for 2-4 weeks using the investigational foot (B) and 2-4 weeks using the usual foot (A2). Outcome is B- A2.
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | -0.2 (11.6)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.798, Wilcoxon signed-rank test

9. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Prosthetic Evaluation Questionnaire (PEQ): Utility Subscale
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | 4.2 (15.4)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.382, Wilcoxon signed-rank test

10. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Prosthetic Evaluation Questionnaire (PEQ): Sound Subscale
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | -8.9 (30.2)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.179, Wilcoxon signed-rank test

11. Secondary Outcome: Difference Between Investigational Foot and Usual Foot in the Comprehensive Lower Extremity Amputee Socket Survey (CLASS): Suspension Subscales
Description: The intent of the CLASS Suspension is to provide greater insight into the cause of socket dissatisfaction compared to the Socket Comfort Score. This subcategory contains 4 items scored using a 5-point scale that relate to common tasks such as standing, sitting, walking, and ascending and descending stairs.
  Scale range: 0-16 Values: 0 = worst outcome; 16 = best outcome
Time Frame: as for outcome 1
Population: All
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lower Extremity Amputees
Number analyzed (Participants) | 31
score on a scale | 0.2 (11.8)
Statistical Analysis 1: Comparison: Lower Extremity Amputees; Test type: Superiority; p = 0.984, Wilcoxon signed-rank test

ADVERSE EVENTS:
Time Frame: 4-8 weeks per individual participant
Arm/Group | Lower Extremity Amputees
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 6/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Extremity Amputees (N=31)
falls - usual foot condition A2 (General disorders) | 3 (3) — Falls while using the participant's usual foot.
falls - investigational foot condition B (General disorders) | 3 (5) — Falls while using the investigational foot.
Residual limb pain usual foot condition A2 (Musculoskeletal and connective tissue disorders) | 0 (0) — Residual limb pain affecting the use of the prosthesis
Residual limb pain investigational foot condition B (Musculoskeletal and connective tissue disorders) | 1 (1) — Residual limb pain affecting the use of the prosthesis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT03703232/Prot_SAP_ICF_000.pdf